CLINICAL TRIAL: NCT00577798
Title: Cardiac MRI for Assessment of Cardiac Structure and Function Following Doxorubicin Based Chemotherapy for Newly Diagnosed Non-Hodgkin's Lymphoma or Hodgkin's Lymphoma
Brief Title: Cardiac Magnetic Resonance Imaging in Patients With Non-Hodgkin Lymphoma or Hodgkin Lymphoma Receiving Doxorubicin
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0409-07-FB; P30CA036727 (NIH); UNMC-40907 (Other Grant/Funding Number: University of Nebraska Medical Center)
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Results first posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Cardiac Toxicity; Chemotherapeutic Agent Toxicity; Lymphoma
Keywords: chemotherapeutic agent toxicity; cardiac toxicity; stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; cutaneous B-cell non-Hodgkin lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; Waldenstrom macroglobulinemia; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult Burkitt lymphoma; stage I adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage I adult lymphoblastic lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; stage I grade 1 follicular lymphoma; stage III grade 1 follicular lymphoma; stage IV grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; stage I grade 2 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; contiguous stage II marginal zone lymphoma; noncontiguous stage II marginal zone lymphoma; stage I marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma
MeSH Terms: conditions — Cardiotoxicity; Lymphoma; Hodgkin Disease; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Only had observational arm
  Interventions: Procedure: contrast-enhanced magnetic resonance imaging

INTERVENTIONS:
Procedure: contrast-enhanced magnetic resonance imaging — Cardiac magnetic resonance imaging (cMRI) offers the unique advantage of being able to analyze both function and structure (myocardial changes in the form of both a functional decrease in ejection fraction and structural changes within the myocardium defined as delayed contrast uptake). Participants will have already received doxorubicin hydrochloride as standard therapy when undergoing chemotherapy for non-Hogdkin's lymphoma and Hogdkin's lymphoma.

SUMMARY:
RATIONALE: Diagnostic procedures, such as cardiac magnetic resonance imaging, may help doctors detect early changes in the heart caused by chemotherapy.

PURPOSE: This clinical trial is studying how well cardiac magnetic resonance imaging works in patients with newly diagnosed non-Hodgkin lymphoma or Hodgkin lymphoma receiving doxorubicin.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether early myocardial structural and functional changes can be detected using cardiac MRI in patients with newly diagnosed non-Hodgkin lymphoma or Hodgkin lymphoma receiving doxorubicin hydrochloride-based chemotherapy.

OUTLINE: Patients undergo cardiac MRI with gadolinium contrast prior to initiation of doxorubicin hydrochloride-based chemotherapy and 3 months after completion of six courses of chemotherapy for non-Hodgkin lymphoma and twelve courses of chemotherapy for Hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-Hodgkin lymphoma or Hodgkin lymphoma

  o Newly diagnosed disease
* Planning to receive doxorubicin hydrochloride-based chemotherapy solely at the University of Nebraska Medical Center
* Fertile patients must use effective contraception
* Able to lie flat for 90 minutes
* Able to fulfill the requirements of the study

Exclusion Criteria:

* Not pregnant or nursing
* No pacemaker
* No chronic kidney disease stages 3-5 (glomerular filtration rate < 60 mL/min)
* No metallic foreign body not approved for MRI
* No known hypersensitivity to gadolinium contrast or other required drugs in the study
* No comorbidity or condition which, in the opinion of the investigator, may interfere with the assessments and procedures of this study
* No prior chemotherapy
* No prior radiotherapy to mantle or mediastinum

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 18 years and above were eligible if they had a new diagnosis (World Health Organization classification) of Non-Hodgkin Lymphoma who planned to undergo doxorubicin-based chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2010-03-01 (Actual); Study Completion 2013-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Porter, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Eppley Cancer Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Lightfoot JC, D'Agostino RB Jr, Hamilton CA, Jordan J, Torti FM, Kock ND, Jordan J, Workman S, Hundley WG. Novel approach to early detection of doxorubicin cardiotoxicity by gadolinium-enhanced cardiovascular magnetic resonance imaging in an experimental model. Circ Cardiovasc Imaging. 2010 Sep;3(5):550-8. doi: 10.1161/CIRCIMAGING.109.918540. Epub 2010 Jul 9. PMID 20622140
- [Background] Kutty S, Rangamani S, Venkataraman J, Li L, Schuster A, Fletcher SE, Danford DA, Beerbaum P. Reduced global longitudinal and radial strain with normal left ventricular ejection fraction late after effective repair of aortic coarctation: a CMR feature tracking study. Int J Cardiovasc Imaging. 2013 Jan;29(1):141-50. doi: 10.1007/s10554-012-0061-1. Epub 2012 May 12. PMID 22581073
- [Background] Poterucha JT, Kutty S, Lindquist RK, Li L, Eidem BW. Changes in left ventricular longitudinal strain with anthracycline chemotherapy in adolescents precede subsequent decreased left ventricular ejection fraction. J Am Soc Echocardiogr. 2012 Jul;25(7):733-40. doi: 10.1016/j.echo.2012.04.007. Epub 2012 May 10. PMID 22578518
- [Background] Sipola P, Vanninen E, Jantunen E, Nousiainen T, Kiviniemi M, Hartikainen J, Kuittinen T. A prospective comparison of cardiac magnetic resonance imaging and radionuclide ventriculography in the assessment of cardiac function in patients treated with anthracycline-based chemotherapy. Nucl Med Commun. 2012 Jan;33(1):51-9. doi: 10.1097/MNM.0b013e32834bfec4. PMID 22044862

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients 18 years and above were eligible if they had a new diagnosis (World Health Organization classification) of Non-Hodgkin's lymphoma (NHL) who planned to undergo doxorubicin-based chemotherapy.
Pre-assignment Details: Patients 18 years and above were eligible if they had a new diagnosis (World Health Organization classification) of NHL who planned to undergo doxorubicin-based chemotherapy.
  Patients were excluded if they had chronic kidney disease grade ≥2, active cardiac disease, or symptoms consistent with congestive heart failure.
Groups:
- Contrast-enhanced Magnetic Resonance Imaging: Doxorubicin hydrochloride: Standard therapy for patients undergoing chemotherapy for their non-Hogdkin's lymphoma and Hogdkin's lymphoma
  Contrast-enhanced magnetic resonance imaging: Cardiac magnetic resonance imaging (cMRI) offers the unique advantage of being able to analyze both function and structure (myocardial changes in the form of both a functional decrease in ejection fraction and structural changes within the myocardium defined as delayed contrast uptake).
Period: Overall Study
Arm/Group | Contrast-enhanced Magnetic Resonance Imaging
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Group: Doxorubicin hydrochloride: Standard therapy for patients undergoing chemotherapy for their non-Hogdkin's lymphoma and Hogdkin's lymphoma
  Contrast-enhanced magnetic resonance imaging: Cardiac magnetic resonance imaging (cMRI) offers the unique advantage of being able to analyze both function and structure (myocardial changes in the form of both a functional decrease in ejection fraction and structural changes within the myocardium defined as delayed contrast uptake).
Arm/Group | Single Group
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 59 [55 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Ejection Fraction (LVEF) and Global Strain Decrease After Doxorubicin Chemotherapy
Description: A reduction of 10% in left ventricular ejection fraction (LVEF) between the two cMRI studies was considered a subclinical functional event. New or progressive myocardial delayed enhancement within ≥1 segment was deemed as a subclinical structural event. Global left ventricle (LV) radial, circumferential, and longitudinal strain data for each patient were compared between cMRI-1 and cMRI-2.
  The study had a fixed endpoint (3 months post-treatment)
Time Frame: cMRI will be done prior to induction of doxorubicin based chemotherapy and at three months after completion of the doxorubicin based chemotherapy regimen.
Population: Ejection fraction (EF) and delayed gadolinium enhancement from cMRI at baseline and 3 months post-treatment will be determined and tested.
Measure: Count of Participants; unit: Participants
Arm/Group | Contrast-enhanced Magnetic Resonance Imaging
Number analyzed (Participants) | 10
Participants
  EF determined from cMRI at baseline and 3 months post-treatment. | 5
  Delayed gadolinium enhancement from cMRI at baseline and 3 months post-treatment. | 5

ADVERSE EVENTS:
Arm/Group | Single Group
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes